CLINICAL TRIAL: NCT00908219
Title: A Prospective, Phase II Trial of Intravenous Bevacizumab (Avastin) for the Prevention of Recurrent Malignant Ascites
Brief Title: A Study of Bevacizumab to Prevent Malignant Ascites
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Accrual closed by sponsor due to lack of accrual and study progress
Sponsor: Baylor College of Medicine (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Martha Mims, Associate Professor, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: H-21728; AVF4534s
Record Dates: First submitted 2009-05-21; First posted 2009-05-25 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2012-02

CONDITIONS: Malignant Ascites
Keywords: malignant ascites; bevacizumab; vascular endothelial growth factor (VEGF); paracentesis
MeSH Terms: interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bevacizumab IV (Experimental): All subjects will be treated with an intravenous infusion of the experimental drug (Bevacizumab 15 mg/kg) every 3 weeks for a total of twelve (12) weeks on study.
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab is given as an IV infusion of 15 mg/kg every three weeks for 12 weeks.
  Other Names: Avastin; RO4876646

SUMMARY:
The purpose of this study is to determine the effectiveness of using Bevacizumab in the prevention of recurrent malignant ascites.

Ascites is a debilitating and unpleasant complication of several types of cancer. Animal and laboratory studies have shown that tumor cell production and/or increases in the amount of Vascular Endothelial Growth Factor (VEGF) is a major cause of the formation of malignant ascites. Therefore, giving patients with malignant ascites a drug that targets and neutralizes VEGF should prevent the recurrence of malignant ascites following paracentesis (a procedure to remove fluid from the abdominal cavity).

DETAILED DESCRIPTION:
All subjects will be treated with an intravenous infusion of the experimental drug (Bevacizumab 15 mg/kg) every 3 weeks for a total of twelve (12) weeks on study. The primary endpoint will be time to the need for repeat abdominal paracentesis after the start of therapy. Secondary endpoints will include an analysis of the mean number of paracenteses required in each subject over the course of 3 months, determination of the repeat paracentesis response rate (proportion of subjects who have a doubling in baseline time to repeat paracentesis) and an assessment of the effect of treatment on quality of life using a subject questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Persistent or symptomatic ascites with positive cytology secondary to any histologically confirmed tumor type not amenable to cytoreductive surgery or additional chemotherapy
* Patients may enroll in this study irrespective of previous therapy including diuretics, surgery, chemotherapy, immunotherapy and radiation therapy
* Must have received a minimum of two paracentesis procedures and a trial of diuretic therapy within 60 days of study entry
* Age Restrictions: 18 years and older
* Life Expectancy: 12 weeks or more
* ECOG Performance Status: 0 -3
* Able and willing to provide informed consent and comply with study and/or follow-up procedures
* Normal organ and marrow function as defined by: Leukocytes >/= 3,000/mcL; Absolute neutrophil count >/= 1,500/mcL; Platelets >/= 100,000/mcL; Total bilirubin within normal institutional limits; AST (SGOT)/ALT(SGPT) </= 2.5 X institutional upper limit of normal (ULN); Creatinine within normal institutional limits OR Creatinine clearance >/+ 60 mL/min for patients with creatinine levels above the institutional normal; Serum Potassium within normal institutional limits; Serum Sodium within normal institutional limits

Exclusion Criteria:

* Patients having received Bevacizumab as part of the treatment of their malignancy within 60 days prior to study entry
* Current, recent (within 30 days of the first infusion of this study) or planned administration of chemotherapy (including all routes of administration), immunotherapy, biologic therapy, radiation therapy or any other anti-VEGF therapy (e.g., tyrosine kinase inhibitors)
* Current, recent (within 30 days of the first infusion of this study), or planned participation in any other experimental drug study
* Pregnant women; A serum pregnancy test will be given to females of childbearing potential prior to study enrollment and the participant must agree to use adequate contraception (barrier or hormonal methods) prior to study entry and for the duration of study participation.
* Un-controlled hypertension (defined as systolic blood pressure > 150 mmHg and/or diastolic blood pressure > 100 mmHg
* History of hypertensive crisis or hypertensive encephalopathy
* New York Heart Association (NYHA) Grade II or greater congestive heart failure
* History of myocardial infarction, unstable angina, stroke or transient ischemic attack within 6 months prior to study entry
* Known CNS disease, except for treated brain metastasis.
* Significant vascular disease (e.g., aortic aneurysm, requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to study entry
* History of hemoptysis (>/= 1/2 teaspoon of bright red blood per episode) within 1 month prior to study entry
* Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation)
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to study entry or anticipation of need for major surgical procedure during the course of the study
* Core biopsy or other minor surgical procedure, excluding placement of a vascular access device or paracentesis/thoracentesis, within 7 days prior to study entry
* History of abdominal fistula or gastrointestinal perforation within 6 months prior to study entry
* Any bowel obstruction that has not fully recovered despite medical or surgical intervention prior to study entry
* Evidence of bowel wall thickening outside the site of the known primary malignancy on baseline radiographs
* Serious, non-healing wound, active ulcer, or untreated bone fracture
* Proteinuria as demonstrated by a Urine Protein/Creatinine ration >/= 1.0 at screening
* Known hypersensitivity to any component of bevacizumab
* Intrathoracic lung carcinoma of squamous cell histology.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-07; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
To determine the repeat paracentesis response rate defined as a doubling of the patient's baseline time to repeat paracentesis. | 12 weeks after initiation of study treatment

SECONDARY OUTCOMES:
To assess the time to the need for the first repeat abdominal paracentesis after the start of Bevacizumab therapy as compared with historical control data. | Unspecified - depends upon when subject will need repeat paracentesis
To analyze the mean number of paracentesis procedures required in each patient over the course of three months. | 12 weeks after the initiation of study treatment
To assess the effect of anti-VEGF therapy on quality of life in patients with malignant ascites. | Every three weeks while on-study

CONTACTS AND LOCATIONS:
Overall Officials: Martha P Mims, MD, PhD, Principal Investigator — Baylor College of Medicine
Locations (3):
- United States (3):
  - Baylor College of Medicine, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - Michael E. DeBakey Veterans Affairs Medical Center, Houston, Texas

REFERENCES:
- [Background] Braunwald, et al. Harrison's Principles of Internal Medicine, 15th Ed. (McGraw-Hill 2001) 517
- [Background] Hurwitz H, Fehrenbacher L, Novotny W, Cartwright T, Hainsworth J, Heim W, Berlin J, Baron A, Griffing S, Holmgren E, Ferrara N, Fyfe G, Rogers B, Ross R, Kabbinavar F. Bevacizumab plus irinotecan, fluorouracil, and leucovorin for metastatic colorectal cancer. N Engl J Med. 2004 Jun 3;350(23):2335-42. doi: 10.1056/NEJMoa032691. PMID 15175435
- [Background] Smith EM, Jayson GC. The current and future management of malignant ascites. Clin Oncol (R Coll Radiol). 2003 Apr;15(2):59-72. doi: 10.1053/clon.2002.0135. PMID 12708713
- [Background] Xu L, Yoneda J, Herrera C, Wood J, Killion JJ, Fidler IJ. Inhibition of malignant ascites and growth of human ovarian carcinoma by oral administration of a potent inhibitor of the vascular endothelial growth factor receptor tyrosine kinases. Int J Oncol. 2000 Mar;16(3):445-54. doi: 10.3892/ijo.16.3.445. PMID 10675474
- [Background] Yukita A, Asano M, Okamoto T, Mizutani S, Suzuki H. Suppression of ascites formation and re-accumulation associated with human ovarian cancer by an anti-VPF monoclonal antibody in vivo. Anticancer Res. 2000 Jan-Feb;20(1A):155-60. PMID 10769648
- [Background] Zebrowski BK, Liu W, Ramirez K, Akagi Y, Mills GB, Ellis LM. Markedly elevated levels of vascular endothelial growth factor in malignant ascites. Ann Surg Oncol. 1999 Jun;6(4):373-8. doi: 10.1007/s10434-999-0373-0. PMID 10379858
- [Background] Verheul HM, Hoekman K, Jorna AS, Smit EF, Pinedo HM. Targeting vascular endothelial growth factor blockade: ascites and pleural effusion formation. Oncologist. 2000;5 Suppl 1:45-50. doi: 10.1634/theoncologist.5-suppl_1-45. PMID 10804091
- [Background] Luo JC, Toyoda M, Shibuya M. Differential inhibition of fluid accumulation and tumor growth in two mouse ascites tumors by an antivascular endothelial growth factor/permeability factor neutralizing antibody. Cancer Res. 1998 Jun 15;58(12):2594-600. PMID 9635584
- [Background] Zebrowski BK, Yano S, Liu W, Shaheen RM, Hicklin DJ, Putnam JB Jr, Ellis LM. Vascular endothelial growth factor levels and induction of permeability in malignant pleural effusions. Clin Cancer Res. 1999 Nov;5(11):3364-8. PMID 10589746
- [Background] Senger DR, Galli SJ, Dvorak AM, Perruzzi CA, Harvey VS, Dvorak HF. Tumor cells secrete a vascular permeability factor that promotes accumulation of ascites fluid. Science. 1983 Feb 25;219(4587):983-5. doi: 10.1126/science.6823562.
- [Background] Numnum TM, Rocconi RP, Whitworth J, Barnes MN. The use of bevacizumab to palliate symptomatic ascites in patients with refractory ovarian carcinoma. Gynecol Oncol. 2006 Sep;102(3):425-8. doi: 10.1016/j.ygyno.2006.05.018. Epub 2006 Jun 23. PMID 16797681
- [Background] Pichelmayer O, Gruenberger B, Zielinski C, Raderer M. Bevacizumab is active in malignant effusion. Ann Oncol. 2006 Dec;17(12):1853. doi: 10.1093/annonc/mdl143. Epub 2006 Jun 21. No abstract available. PMID 16790519
- [Background] Ozcan C, Wong SJ, Hari P. Reversible posterior leukoencephalopathy syndrome and bevacizumab. N Engl J Med. 2006 Mar 2;354(9):980-2; discussion 980-2. No abstract available. PMID 16514715
- [Background] Scappaticci FA, Fehrenbacher L, Cartwright T, Hainsworth JD, Heim W, Berlin J, Kabbinavar F, Novotny W, Sarkar S, Hurwitz H. Surgical wound healing complications in metastatic colorectal cancer patients treated with bevacizumab. J Surg Oncol. 2005 Sep 1;91(3):173-80. doi: 10.1002/jso.20301. PMID 16118771
- [Background] Sandler A, Gray R, Perry MC, Brahmer J, Schiller JH, Dowlati A, Lilenbaum R, Johnson DH. Paclitaxel-carboplatin alone or with bevacizumab for non-small-cell lung cancer. N Engl J Med. 2006 Dec 14;355(24):2542-50. doi: 10.1056/NEJMoa061884. PMID 17167137
- [Background] Miller KD, Chap LI, Holmes FA, Cobleigh MA, Marcom PK, Fehrenbacher L, Dickler M, Overmoyer BA, Reimann JD, Sing AP, Langmuir V, Rugo HS. Randomized phase III trial of capecitabine compared with bevacizumab plus capecitabine in patients with previously treated metastatic breast cancer. J Clin Oncol. 2005 Feb 1;23(4):792-9. doi: 10.1200/JCO.2005.05.098. PMID 15681523
- [Background] Karp JE, Gojo I, Pili R, Gocke CD, Greer J, Guo C, Qian D, Morris L, Tidwell M, Chen H, Zwiebel J. Targeting vascular endothelial growth factor for relapsed and refractory adult acute myelogenous leukemias: therapy with sequential 1-beta-d-arabinofuranosylcytosine, mitoxantrone, and bevacizumab. Clin Cancer Res. 2004 Jun 1;10(11):3577-85. doi: 10.1158/1078-0432.CCR-03-0627. PMID 15173063
- [Background] Wedam SB, Low JA, Yang SX, Chow CK, Choyke P, Danforth D, Hewitt SM, Berman A, Steinberg SM, Liewehr DJ, Plehn J, Doshi A, Thomasson D, McCarthy N, Koeppen H, Sherman M, Zujewski J, Camphausen K, Chen H, Swain SM. Antiangiogenic and antitumor effects of bevacizumab in patients with inflammatory and locally advanced breast cancer. J Clin Oncol. 2006 Feb 10;24(5):769-77. doi: 10.1200/JCO.2005.03.4645. Epub 2006 Jan 3. PMID 16391297
- [Background] D'Adamo DR, Anderson SE, Albritton K, Yamada J, Riedel E, Scheu K, Schwartz GK, Chen H, Maki RG. Phase II study of doxorubicin and bevacizumab for patients with metastatic soft-tissue sarcomas. J Clin Oncol. 2005 Oct 1;23(28):7135-42. doi: 10.1200/JCO.2005.16.139. PMID 16192597